CLINICAL TRIAL: NCT00964860
Title: A Controlled Clinical Study to Determine the Gingivitis Benefit of Flossing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009061
Record Dates: First submitted 2009-08-20; First posted 2009-08-25 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brushing Only (No Intervention): Brushing Only with an Oral B manual toothbrush and Crest Cavity Protection, sodium fluoride dentifrice
- Brushing + Flossing (Experimental): Brushing with an Oral B manual toothbrush and Crest Cavity Protection, sodium fluoride dentifrice, plus flossing with Glide floss
  Interventions: Device: Glide dental floss

INTERVENTIONS:
Device: Glide dental floss — Glide waxed dental floss
  Arms: Brushing + Flossing

SUMMARY:
This is a randomized, controlled, examiner-blind, parallel group, four week clinical study comparing brushing plus flossing to brushing alone in 60 healthy adults with pre-existing gingivitis.

ELIGIBILITY:
Inclusion Criteria:

In order to be included in the study, each subject must:

* be at least 18 years of age;
* be physically able to floss their teeth;
* have a minimum of 18 natural teeth (teeth that are grossly carious, fully crowned, or extensively restored will not be included);
* have refrained from performing oral hygiene the morning of the Baseline visit;
* be in good general health;
* have interproximal MGI (Modified Gingival Index) score of >2.8.

Exclusion Criteria:

Subjects are excluded from study participation where there is evidence of:

* severe periodontal disease;
* discoloration or pigmentation in the gingival tissue;
* meaningful misalignment of front teeth;
* fixed facial orthodontic appliances;
* use of antibiotics within two weeks of the Baseline Visit and at any time during the study;
* any diseases or conditions that could be expected to interfere with the subject safely completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Witt, PhD, Study Director — Procter and Gamble
Locations (1):
- Radiologio Oral Y Maxilofacial, Guatemala City, Guatemala

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brushing Only | Brushing + Flossing
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brushing Only | Brushing + Flossing | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.0 (7.8) | 28.2 (8.5) | 28.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  Guatemala | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Interproximal Lobene Modified Gingival Index Between the Brushing Only Group and the Brushing + Flossing Group
Description: Gingivitis was scored using the Lobene Modified Gingival Index (a visual examination for inflammation) on all scorable teeth. For each tooth, six gingival areas (distobuccal, buccal, mesiobuccal, mesiolingual, lingual, and distolingual) were scored on a 5-point, categorical scale (0 = absence of inflammation; 4 = severe inflammation) corresponding to Inflammation
Time Frame: 30 days
Population: per protocol
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brushing Only | Brushing + Flossing
Number analyzed (Participants) | 30 | 29
units on a scale | 2.11 (0.05) | 1.87 (0.05)
Statistical Analysis 1: Comparison: Brushing Only vs Brushing + Flossing; Test type: Superiority or Other; p = 0.001, ANCOVA — a priori threshold for statistical significance = 0.05; Mean Difference (Final Values) = 0.24, Standard Error of Mean 0.05 — All treatment comparisons were 1-sided with the significance level set at 5%. Units on the MGI Scale

2. Secondary Outcome: Whole Mouth Mean Lobene Modified Gingival Index Between the Brushing Only Group and the Brushing + Flossing Group
Description: Whole-mouth average MGI scores were calculated separately for each subject and visit by averaging the MGI scores of all gradable sites. Interpoximal average MGI scores were also calculated for each subject and visit by averaging over only interpoximal sites (buccal-mesial, buccal-distal, lingual-mesian, and lingual-distal).
  Within each treatment, changes from baseline were analyzed using paired t-test. Between treatments mean comparisons were conducted using analysis of covariance with baseline MGI score as a covariate. All statistical comparisons were two-sided with a 5% significance level.
  The average MGI score for a subject can range from 0 (no gingivitis) to 4 (inflammation on all gradable sites).
Time Frame: 30 days
Population: per protocol
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brushing Only | Brushing + Flossing
Number analyzed (Participants) | 30 | 29
units on a scale | 2.06 (0.05) | 1.86 (0.05)
Statistical Analysis 1: Comparison: Brushing Only vs Brushing + Flossing; Test type: Superiority or Other; p = 0.004, ANCOVA — a priori threshold for statistical significance = 0.05; Mean Difference (Final Values) = 0.20, Standard Error of Mean 0.05 — All treatment comparisons were 1-sided with the significance level set at 5%

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Brushing Only | Brushing + Flossing
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less